CLINICAL TRIAL: NCT00218517
Title: Selegiline for Treatment of Cannabis Dependence
Brief Title: Effectiveness of Selegiline in Treating Marijuana Dependent Individuals - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Ivan Montoya, Program Official, NIDA
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-19246-1; R21-19246-1; DPMC
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-09

CONDITIONS: Marijuana Abuse
Keywords: cannabis use disorder
MeSH Terms: conditions — Marijuana Abuse | interventions — Selegiline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Selegiline hydrochloride
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Selegiline hydrochloride — Daily oral selegiline, 5 mg po qd x 7 days, then 5 mg po bid for 7 weeks
  Other Names: Selegiline, Selegiline hydrochloride, l-Deprenyl
  Arms: 1
Drug: Placebo — Matching placebo capsules using blue 00 capsules
  Arms: 2

SUMMARY:
During the past 15 years, the demand for treatment for marijuana-related problems in the United States has increased nearly twofold. Selegiline is a medication currently used to treat nicotine dependence. The purpose of this study is to evaluate whether selegiline may be useful in treating individuals with marijuana dependence.

DETAILED DESCRIPTION:
Behavioral therapy paired with drug therapy might be a more effective treatment approach to marijuana dependence than behavioral therapy alone. Selegiline is a monoamine oxidase-B inhibitor. It increases dopamine activity in parts of the brain that are involved in dependence on addictive drugs such as nicotine, cocaine, and marijuana. Selegiline has been effective in treating nicotine dependence, but has not yet been studied in treating marijuana dependent individuals. The purpose of this study is to evaluate the effectiveness of selegiline in treating marijuana dependent individuals. Specifically, this study will determine whether selegiline reduces marijuana craving and withdrawal symptoms, thus leading to reduction or abstinence in marijuana use.

Participants in this 9-week, double-blind, placebo-controlled study will be randomly assigned to receive either selegiline (10 mg/day in two 5 mg pills) or placebo. Study visits will occur twice each week. At each study visit, participants will complete self-reports and urine toxicology tests. Throughout the study, participants will receive weekly individual counseling. The counseling sessions will last 15 minutes. Reduction in marijuana use as well as the number of weeks of consecutive marijuana abstinence will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for current marijuana dependence
* Positive urine toxicology test for marijuana
* Reports current marijuana use
* Weighs at least 100 lbs
* Women of childbearing age will be included provided they agree to use adequate contraception

Exclusion Criteria:

* Meets dependence or abuse criteria for alcohol
* Meets dependence criteria for illicit substances other than marijuana
* Serious medical disorders (such as unstable angina or liver failure), that may make participation in the trial unsafe
* Pregnant
* Currently diagnosed with a psychotic disorder
* Currently suicidal or pose a homicidal risk
* Currently taking over-the-counter (e.g., pseudoephedrine) or prescription (e.g., methylphenidate) sympathomimetic agents, antidepressant agents (e.g., tricyclic antidepressants, serotonin reuptake inhibitors, bupropion, other monoamine oxidase inhibitors), or meperidine (Demerol)
* Unable to understand English
* Known hypersensitivity to selegiline hydrochloride

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2005-03; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Marijuana addiction severity, Week 9
Marijuana withdrawl symptoms, Week 9

CONTACTS AND LOCATIONS:
Overall Officials: Brent A Moore, Ph.D., Principal Investigator — Yale University
Locations (1):
- MRU, New Haven, Connecticut, United States